CLINICAL TRIAL: NCT00731042
Title: A Two-week Crossover Evaluation of Two Hand Antiseptic Products on Skin Condition in Healthy Human Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: I2MS05-010877
Record Dates: First submitted 2008-08-06; First posted 2008-08-08 (Estimated); Results first posted 2009-06-17 (Estimated); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Healthy
Keywords: Skin health
MeSH Terms: interventions — chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Avagard (Experimental): 3M Avagard Surgical and healthcare Personnel Hand Antiseptic with Moisturizers
  Interventions: Drug: Avagard
- Purell (Active Comparator): Purell Surgical Scrub with Moisturizers
  Interventions: Drug: Purell Surgical Scrub

INTERVENTIONS:
Drug: Avagard — Topical solution, 6 mL, 6 applications/day for 14 days.
  Arms: Avagard
Drug: Purell Surgical Scrub — Topical solution, 4 mL, 6 applications/day for 14 days.
  Other Names: Purell Surgical Scrub with Moisturizers
  Arms: Purell

SUMMARY:
Evaluate the effect of two hand antiseptic products on hand skin conditions of healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Female age 25 - 55
* Subject agrees not to use any hand wash products on their hands other than what has been provided in the study.
* Subject agrees not to use any moisturizers or any skin products on their hands during the study
* Subject agrees to use gloves to protect hands from activities such as dish washing
* Subject is willing to sign the Informed Consent and HIPAA
* Subject agrees to comply with the study requirement

Exclusion Criteria:

* Subject has a history of psoriasis, active dermatitis, skin reactions, cracked, irritated, broken skin, skin infection on their hands
* Subject has scaly skin on hands based on Visual Scoring Scale at Day 1
* Subject has a sensitivity or history of skin reactions to any study materials (eg, alcohol, chlorhexidine gluconate or zinc pyrithone or latex in the gloves)
* Subject has been using moisturizing products or any products on their arms and hands within 5 days prior to participation in the study
* Subject is pregnant
* Study coordinator believes the subject is unsuitable for inclusion in the study

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2008-03; Primary Completion 2008-04 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary L Grove, PhD, Principal Investigator — cyberDERM Clinical Research

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After screening, there was a 5-days washout prior to enrollment into period 1. This was then followed by another 5-days washout between periods 1 and 2.
Groups:
- Purell First Followed by Avagard: Using Purell for 14 days. Rest for 5 days(no product used). Then use Avagard for 14 days.
- Avagard First Followed by Purell: Using Avagard for 14 days. Rest for 5 days(no product used). Then use Purell for 14 days.
Period: First Intervention
Arm/Group | Purell First Followed by Avagard | Avagard First Followed by Purell
Started | 16 | 17
Completed | 16 | 17
Not Completed | 0 | 0
Period: Wash-out
Arm/Group | Purell First Followed by Avagard | Avagard First Followed by Purell
Started | 16 | 17
Completed | 16 | 17
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Purell First Followed by Avagard | Avagard First Followed by Purell
Started | 16 | 17
Completed | 16 | 15 (2 subjects did not met inclusion criteria for Period 2 Visual scoring skin condition)
Not Completed | 0 | 2
Not completed — Did not meet inclusion criteria | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Purell First Followed by Avagard | Avagard First Followed by Purell | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 17 | 33
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 33
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Skin Health, Visual Skin Score (VSS) at 14 Days
Description: Observe VSS score at 14 days, and graded change of skin health from baseline using scale of 0 (normal) - 5 (very scaly).
Time Frame: Baseline and 14 days
Population: Analysis was done per protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Purell First Followed by Avagard | Avagard First Followed by Purell
Number analyzed (Participants) | 15 | 15
units on a scale | 0.1 (1.11) | 0.4 (1.53)

ADVERSE EVENTS:
Description: The number of participants affected/at risk in the adverse event reporting section was recorded as "0". Adverse events and Serious adverse events were collected and assessed, but none observed.
Arm/Group | Purell First Followed by Avagard | Avagard First Followed by Purell
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 0/16 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI was a test lab, and they do not publish study result. Sponsor can choose to publish.